CLINICAL TRIAL: NCT05612854
Title: Catheter Directed Therapy for Intermediate Risk Pulmonary Embolism Patients Guided by Prediction Model for Impending Shock
Brief Title: Catheter Directed Therapy in Intermediate Risk Pulmonary Embolism Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayman khairy Mohamed, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDT in pulmonary embolism
Record Dates: First submitted 2022-10-16; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Pulmonary Embolism Subacute Massive
Keywords: catheter directed therapy; intermediate risk pulmonary embolism

STUDY DESIGN:
Intervention Model Description: Randomized controlled, open-label, parallel-assignment, prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- catheter directed therapy group in intermediate risk pulmonary embolism patients (Active Comparator): in this arm, intermediated risk pulmonary embolism patients is treated by intervention in the form of:
  * A. Mechanical embolectomy: by hydromechanical defragmentation by pigta
  * B. Suction embolectomy: using The Penumbra Indigo aspiration system
  * C. Catheter directed thrombolysis:
  Interventions: Procedure: Mechanical embolectomy: by hydromechanical defragmentation by pigtail; Device: Suction embolectomy by the Penumbra Indigo aspiration system
- medical therapy group in intermediate risk pulmonary embolism patients (Active Comparator): in this arm, intermediated risk pulmonary embolism patients is treated by routine anticoagulation only.
  Interventions: Procedure: Mechanical embolectomy: by hydromechanical defragmentation by pigtail; Device: Suction embolectomy by the Penumbra Indigo aspiration system

INTERVENTIONS:
Procedure: Mechanical embolectomy: by hydromechanical defragmentation by pigtail — Hydro-mechanical defragmentation (HMD) is one of the CDT modalities for high-risk PE patients, in which rapid pigtail rotation is combined with heparinized saline injection for thrombus fragmentation
Device: Suction embolectomy by the Penumbra Indigo aspiration system — The Penumbra Indigo aspiration system (Penumbra Inc., Alameda, CA, USA) that will be used, is an 8-Fr device and its associated tubing, pump, and separator, has the flexibility for placement in segmental branches of the pulmonary arteries.
  510(k) Number :K160449 FOIA Releasable 510(k) K160449 Device Name:Penumbra System, Penumbra Pump MAX

SUMMARY:
Aim of the work:

1. To compare conventional medical therapy versus catheter-directed therapy in intermediate high risk acute pulmonary embolism.
2. To define predictors of progression from intermediate to high-risk in medically-treated patients for ideal timing for intervention.

DETAILED DESCRIPTION:
Based on history, physical examination, surface 12-lead ECG, bed-side echocardiography, patients with a high probability of acute pulmonary embolism are selected and subjected to CT pulmonary angiography to confirm the diagnosis and calculate the pulmonary artery obstruction score.

Routine labs are withdrawn, including cardiac troponin.Methods:

Detailed TTE will be done with emphasis on the following indicators of RV strain and/or dysfunction:

1. Echocardiography findings that are indicative of RV dysfunction

   * tricuspid annular plane systolic excursion (TAPSE)
   * S' Velocity
   * the McConnell's sign
2. RV dilation
3. interventricular septal flattening.
4. elevated right ventricular pressures
5. plethoric inferior vena cava
6. tricuspid regurgitation
7. Direct visualization of thromboembolic in the RT heart and PA
8. RV stroke volume measured by RVOT VTI.
9. LV stroke volume measured by LVOT VTI Intermediate-high risk patient will be identified (based on the calculated pulmonary embolism severity index, RV dysfunction on TTE and/or CT, cardiac troponin), and then randomized to either receiving conventional medical treatment or catheter-directed interventional therapy if the patient consents.

7. Catheter directed therapy

A. Mechanical embolectomy:

Mechanical fragmentation will be done using a 6 F pigtail catheter inserted inside the thrombus guided by the CTPA images.

Hydro-mechanical defragmentation (HMD) is one of the CDT modalities for high-risk PE patients, in which rapid pigtail rotation is combined with heparinized saline injection for thrombus fragmentation.(4)

B. Suction embolectomy:

Suction embolectomy was one of the earliest techniques for transcatheter treatment of PE, and was introduced by Greenfield et al, using a 12-Fr catheter with a cup on its distal end. Suction was applied manually to the catheter hub with a large syringe. (13) The Penumbra Indigo aspiration system (Penumbra Inc., Alameda, CA, USA) that will be used, is an 8-Fr device and its associated tubing, pump, and separator, has the flexibility for placement in segmental branches of the pulmonary arteries. The Indigo aspiration system is indicated for use in the peripheral arterial system and the pulmonary arteries, receiving U.S. Food and Drug Administration 510(k) clearance for PE in December 2019.(14)

C. Catheter directed thrombolysis:

Catheter-directed thrombolysis allows delivery of the thrombolytic agent directly to the area of highest embolic burden via a catheter.

Intermediate-high risk patient will be identified (based on the calculated pulmonary embolism severity index, RV dysfunction on TTE and/or CT, cardiac troponin), and then randomized to either receiving conventional medical treatment or catheter-directed interventional therapy if the patient consents.

ELIGIBILITY:
Inclusion Criteria:

* Acute pulmonary embolism patients (confirmed by CT pulmonary angiography [CTPA])
* symptoms started within 15 days of enrollment
* intermediate-high risk pulmonary embolism patients , i.e., who have all of the following risk indicators combined :(2) i.Pulmonary Embolism Severity Index (PESI) class III-V or sPESI ≥1, ii.AND RV dysfunction on TTE or CTPA, iii.AND elevated cardiac troponin levels
* with none of the following high-risk presentations: cardiac arrest, systolic blood pressure <90 mmHg, or vasopressors required to achieve a BP ≥90 mmHg despite an adequate filling status, or end-organ hypoperfusion.

Exclusion Criteria:

* high risk patients who are hemodynamically unstable (cardiogenic shock, SBP <90 mmHg, or use of intotropic support).
* low risk patients with no RV dysfunction.
* Patients with history of CTEPH (or previous acute PE)
* Patients known to have other pulmonary hypertension, apart from group IV (CTEPH).
* Patients with sever kidney injury (eGFR <30 mg/dl/1.7m2).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
1.comparison between conventional medical therapy and catheter-directed therapy in intermediate high risk acute pulmonary embolism patients | up to 2 years
  comparison in intermediate high risk acute pulmonary embolism patients between conventional medical therapy and catheter-directed therapy as regarding safety and efficacy of the therapy by clinical assessment of occurrence of major adverse cardiac events.
1.comparison between conventional medical therapy and catheter-directed therapy in intermediate high risk acute pulmonary embolism patients | up to 2 years
  comparison in intermediate high risk acute pulmonary embolism patients between conventional medical therapy and catheter-directed therapy as regarding safety and efficacy of the therapy by echocardiographic assessment of right ventricular function by TAPSE (mm) , RV/LV diameter ratio ,TR peak gradient (mmHg)
1.comparison between conventional medical therapy and catheter-directed therapy in intermediate high risk acute pulmonary embolism patients | up to 2 years
  comparison in intermediate high risk acute pulmonary embolism patients between conventional medical therapy and catheter-directed therapy as regarding safety and efficacy of the therapy by CT pulmonary angiography to asses embolus size and Pulmonary artery obstruction index

SECONDARY OUTCOMES:
predictors of progression from intermediate to high-risk acute pulmonary embolism patients | up to 2 years
  identifying predictors for ideal timing for intervention in intermediate risk pulmonary embolism patients who are medically-treated by new echocardiographic parameters (LVOT velocity time integral and RVOT velocity time integral)

OTHER OUTCOMES:
Implementation of pulmonary embolism response team at Assiut university hospitals | up to 2 years
  institutional reconstruction and communication between different departments (chest, cardiology, radiology and clinical pathology departments) aiming to implement a pulmonary embolism response team with clear structure and operational levels for decision making

CONTACTS AND LOCATIONS:
Overall Officials: Shrouk K Ali, MSc, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Giri J, Sista AK, Weinberg I, Kearon C, Kumbhani DJ, Desai ND, Piazza G, Gladwin MT, Chatterjee S, Kobayashi T, Kabrhel C, Barnes GD. Interventional Therapies for Acute Pulmonary Embolism: Current Status and Principles for the Development of Novel Evidence: A Scientific Statement From the American Heart Association. Circulation. 2019 Nov 12;140(20):e774-e801. doi: 10.1161/CIR.0000000000000707. Epub 2019 Oct 4. PMID 31585051
- [Background] Hassan AKM, Ahmed H, Ahmed Y, Elfadl AA, Omar A. Efficacy and safety of hydro-mechanical defragmentation in intermediate- and high-risk pulmonary embolism. Egypt Heart J. 2021 Sep 25;73(1):84. doi: 10.1186/s43044-021-00204-2. PMID 34564780
- [Background] Kroupa J, Buk M, Weichet J, Malikova H, Bartova L, Linkova H, Ionita O, Kozel M, Motovska Z, Kocka V. A pilot randomised trial of catheter-directed thrombolysis or standard anticoagulation for patients with intermediate-high risk acute pulmonary embolism. EuroIntervention. 2022 Oct 7;18(8):e639-e646. doi: 10.4244/EIJ-D-21-01080. PMID 35620984